CLINICAL TRIAL: NCT02730858
Title: A Collaborative Palliative and Oncology Care Model for Metastatic Breast Cancer
Brief Title: Palliative and Oncology Care Model in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-585
Record Dates: First submitted 2016-03-24; First posted 2016-04-07 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Palliative Care; Breast Cancer; End of life; Health service research
MeSH Terms: conditions — Breast Neoplasms; Death | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative and oncology care model (Experimental): After the screening procedure confirm eligibility to participate in the research study. Participants will be randomized into one of two study groups;
  -- Standard oncology care with palliative care.
  Interventions: Behavioral: Palliative and Oncology Care
- Standard oncology care (Active Comparator): After the screening procedure confirm eligibility to participate in the research study. Participants will be randomized into one of two study groups;
  -- Standard oncology care
  Interventions: Behavioral: Standard Oncology Care

INTERVENTIONS:
Behavioral: Palliative and Oncology Care — Patients randomized to the intervention will receive collaborative care from palliative care and oncology for the remainder of their illness. The initial five visits with palliative care will be conducted in accordance with the study specific clinical practice guidelines and occur at least monthly.
  Arms: Palliative and oncology care model
Behavioral: Standard Oncology Care — Patients randomized to oncology care alone will continue to receive routine care identical to what they would have received if they had not participated in the trial. Either patients or their oncologists can request palliative care consultation at any point in time.
  Arms: Standard oncology care

SUMMARY:
The purpose of this research study is to test a new way to deliver oncology and palliative care for patients with metastatic breast cancer.

* The goal of this study is to test a model where oncology and palliative care work together to care for participants with metastatic breast cancer who were recently admitted to the hospital or have new or worsening cancer involving their brain or the fluid around the brain or spinal cord.
* The investigators are studying whether participants who receive care from both teams have better communication about their care and improved quality of life and mood compared to those receiving care from only their oncologists.

The purpose of this randomized clinical trial is to conduct a randomized trial testing the impact of the collaborative palliative and oncology care model or standard oncology care models among patients with poor prognosis metastatic breast cancer. Participants assigned to the intervention arm will participate in a series of structured palliative care visits, following tailored clinical practice guidelines previously developed for patients with metastatic breast cancer.

DETAILED DESCRIPTION:
This research study tests whether or not the earlier introduction of a team of clinicians that specialize in the lessening (palliation) of symptoms and addressing quality of life concerns may improve the end-of-life care, quality of life, and mood of women with poor prognosis metastatic breast cancer.

Palliative care is a specific type of medical care given to patients to improve their pain and other symptoms like fatigue, and to support patients and their families as they cope with their illness. Palliative care includes physicians and advanced practice nurses who have been specifically trained in how to help patients with serious illness.

Increasingly, the role of palliative care has been shown to benefit patients when introduced early in the disease trajectory. For example, in patients with metastatic (or spread) lung cancer, early involvement of palliative care improves patients' quality of life and mood. Patients with some metastatic cancers, like breast cancer, have an unpredictable disease trajectory, which makes it difficult to determine the best time to introduce palliative care services.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with metastatic breast cancer and:

  1. have been informed of a diagnosis of leptomeningeal disease in the past eight weeks; OR
  2. have been informed of a diagnosis of progressive brain metastases after initial radiation therapy in the past eight weeks; OR
  3. have been diagnosed brain metastases and began whole brain radiation in the past eight weeks; OR
  4. had an unplanned hospital admission and was discharged within the past eight weeks; OR
  5. have been diagnosed with triple negative breast cancer and started second-line treatment in the past eight weeks; OR
  6. have started the third regimen in one year within the past eight weeks; OR
  7. have HER2+ disease and started third-line therapy within the past eight weeks; OR
  8. have ER+ disease and started third-line chemotherapy within the past eight weeks; OR
  9. enrolled on a clinical trial within the past eight weeks
* Receiving cancer care at MGH Cancer Center.
* Able to read and write in English.
* Eastern Cooperative Oncology Group status between 0 and 2.

Exclusion Criteria:

* Already receiving palliative care in the outpatient setting.
* Active, untreated, unstable, serious mental illness (e.g., active, untreated psychotic, bi-polar, or substance-dependence disorder) interfering with ability to participate.
* Cognitive impairment (e.g., delirium, dementia) interfering with ability to participate.
* Requires urgent palliative or hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05; Primary Completion 2019-09 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
End of life care preference documentation | 1 year
  Compare differences in rate of documentation of end of life care preferences (Yes documented vs. No)

SECONDARY OUTCOMES:
Patient-reported end of life care conversation | 6 months
  Examine patient report of end of life care preferences with their clinician using the following item: "have you and your doctors discussed any particular wishes you have about the care you want to receive if you were dying?" Although patients complete this measure repeatedly during the course of the study, the investigators will use the final assessment either prior to death or at six months follow-up (whichever comes first) for this analysis.
Patient-reported quality of life (FACT-Breast) | Weeks 6, 12, 18, and 24
  Compare patient-reported quality of life between the two study arms at weeks 6, 12, 18, and 24.
Patient-reported depression symptoms (Hospital Anxiety and Depression Scale) | Weeks 6, 12, 18, and 24
  Compare patient-reported depression symptoms between the two study arms at weeks 6, 12, 18, and 24.
Patient-reported anxiety symptoms (Hospital Anxiety and Depression Scale) | Weeks 6, 12, 18, and 24
  Compare patient-reported anxiety symptoms between the two study arms at weeks 6, 12, 18, and 24.
Chemotherapy at the end of life | 14, 7 and 3 days before death
  Examine differences in rates of chemotherapy administration during the last 3, 7, and 14 days of life between the two study arms
Rate of hospice utilization at the end of life | 6 months
  Examine difference the in rates of hospice utilization between the two study arms.
Length of stay on hospice | 6 months
  Examine difference in hospice length-of-stay between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350
- [Derived] Greer JA, Moy B, El-Jawahri A, Jackson VA, Kamdar M, Jacobsen J, Lindvall C, Shin JA, Rinaldi S, Carlson HA, Sousa A, Gallagher ER, Li Z, Moran S, Ruddy M, Anand MV, Carp JE, Temel JS. Randomized Trial of a Palliative Care Intervention to Improve End-of-Life Care Discussions in Patients With Metastatic Breast Cancer. J Natl Compr Canc Netw. 2022 Feb;20(2):136-143. doi: 10.6004/jnccn.2021.7040. PMID 35130492